CLINICAL TRIAL: NCT04125602
Title: Westlake Personalized Nutrition Intervention Study: N-of-1 Trials for Dietary Macronutrient Intake
Brief Title: Westlake N-of-1 Trials for Macronutrient Intake
Acronym: WE-MACNUTR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Westlake University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 20190919ZJS001
Record Dates: First submitted 2019-10-10; First posted 2019-10-14 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2019-10

CONDITIONS: Postprandial Hyperglycemia; Metabolic Disorder, Glucose
Keywords: Personalized Nutrition; Glucose Metabolism; Gut Microbiota
MeSH Terms: conditions — Hyperglycemia; Glucose Metabolism Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High fat low carbohydrate diet (Experimental)
  Interventions: Other: High fat low carbohydrate diet; Other: Low fat high carbohydrate diet
- Low fat high carbohydrate diet (Experimental)
  Interventions: Other: High fat low carbohydrate diet; Other: Low fat high carbohydrate diet

INTERVENTIONS:
Other: High fat low carbohydrate diet — Throughout the 6-day intervention, participants are provided with a high fat, low carbohydrate diet (HF-LCD), including a 3-day diet in which the percentage of fat, protein and carbohydrate is 60%, 15% and 25% respectively while the three macronutrients in the other 3-day diet account for 70%, 15% and 15% respectively. The sequencing of the two diets will be randomized.
  Other Names: HF-LCD
Other: Low fat high carbohydrate diet — Throughout the 6-day intervention, participants are provided with a low fat, high carbohydrate diet (LF-HCD), including a 3-day diet in which the percentage of fat, protein and carbohydrate is 20%, 15% and 65% respectively while the three macronutrients in the other 3-day diet account for 10%, 15% and 75% respectively. The sequencing of the two diets will be randomized.
  Other Names: LF-HCD

SUMMARY:
This is a dietary intervention study in students and staff of Westlake University, which is designed to provide evidence in support of N-of-1 methods as an approach to advance personalized nutrition. The primary aim is using a series of N-of-1 trials to determine the impacts of a high fat, low carbohydrate diet (HF-LC) on glucose metabolism and gut microbiota in subjects versus a low fat, high carbohydrate diet (LF-HC) at both the individual and group level.

DETAILED DESCRIPTION:
This study will employ a series of individual N-of-1 trials comparing a high fat, low carbohydrate diet (HF-LC) to a low fat, high carbohydrate diet (LF-HC). Participants will enter the study on a usual diet and will have a 6-day run in period for diet planning and baseline data collection before beginning their intervention. The HF-LC or the LF-HC will be randomized as the starting intervention followed by a wash-out period lasting for 6 days with normal diet between two interventions to eliminate previous intervention effects. Then the participants will be provided with the other diet. Both HF-LC and LF-HC last for 6 days in each set which consists of two wash-out periods and two intervention periods. There will be 3 sets in this study and investigators will aggregate the results of the completed N-of-1 trials across all participants to estimate the group level impacts of HF-LC compared to LF-HC.

ELIGIBILITY:
Inclusion Criteria:

* Willingness and capability to complete the study protocol

Exclusion Criteria:

* Inability or unwillingness to approved to provide informed consent
* Neurological conditions that might affect the assessment of the study measurement
* Hospitalization or surgery planned within 3 months
* Gastrointestinal diseases
* Other serious medical conditions, such as liver, kidney, or systemic disease
* Women who are pregnant or lactating
* Tobacco, alcohol, or illicit drug abuse
* Had taken antibiotics in the past two weeks prior to the start of the trial
* Participants on a vegan diet
* Any food allergy
* Lack of smart phone and data plan for participating caregiver
* Non-Chinese speaking participants
* Participating in another concurrent intervention study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-10-20 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Postprandial blood glucose change | Day 7-12 and day 19-24 of each set
  Postprandial blood glucose from different foods will be assessed.
Blood glucose profiling | Day 7-12 and day 19-24 of each set
  Glucose levels will be recorded by continuous glucose monitoring over the intervention periods.

OTHER OUTCOMES:
Fecal metabolites | Day 1, day7, day 13 and day 19 of each set
  Fecal metabolite extracts will be analysed by performing liquid chromatography/quadrupole time-of-flight mass spectrometry (LC/Q-TOF/MS).
Fecal microbiota | Day 1, day7, day 13 and day 19 of each set
  Gut microbial communities and their abundant features will be analysed based on shotgun metagenomic sequencing.
Metabolomics profiling | Day 1, day7, day 13 and day 19 of each set
  Targeted metabonomics are analyzed based on urine and faeces at all visits (also based on serum in set 1).
Laboratory markers of glucose metabolism and inflammation | Day 1, day7, day 13 and day 19 of set 1
  insulin, leptin, adiponection, free fatty acid, Interleukin(IL)-6, IL-8, IL-10, IL-12, IL-17A, IL-1ra, tumour necrosis factor alpha (TNF-α), Lipopolysaccharide binding protein (LBP), cortisol, high-sensitivity C-reactive protein, serum amyloid A, soluble E-selectine, soluble intracellular adhesion molecule-1, plasminogen activator inhibitor-1, vascular cell adhesion molecule, monocyte chemoattractant protein (MCP)-1, adrenaline, noradrenaline, peptide YY, and neuropeptide Y are tested at all visits of set 1.
Lipid metabolism | Day 1, day7, day 13 and day 19 of set 1
  Triglyceride, cholesterol, high density lipoprotein cholesterol, low density lipoprotein cholesterol, apolipoprotein A1 and apolipoprotein B are tested at all visits of set 1.
Physiological characteristics | Day 1, day7, day 13 and day 19 of set 3
  Weight and blood pressure are collected at all visits of set 3.

CONTACTS AND LOCATIONS:
Overall Officials: Ju-Sheng Zheng, PhD, Principal Investigator — Westlake University
Locations (1):
- Westlake University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tian Y, Ma Y, Fu Y, Zheng JS. Application of n-of-1 Clinical Trials in Personalized Nutrition Research: A Trial Protocol for Westlake N-of-1 Trials for Macronutrient Intake (WE-MACNUTR). Curr Dev Nutr. 2020 Aug 26;4(9):nzaa143. doi: 10.1093/cdn/nzaa143. eCollection 2020 Sep. PMID 32968703